CLINICAL TRIAL: NCT01535612
Title: A Study Evaluating the Feasibility of Use and Performance of PaQ™ in Patients With Type 2 Diabetes Mellitus Who Are Currently Treated With Basal/Bolus Insulin Therapy
Brief Title: Study of PaQ™ (a Simple Patch on Insulin Delivery Device) in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CeQur Corporation (Industry)
Collaborators: International Diabetes Center at Park Nicollet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQR-09001
Record Dates: First submitted 2011-09-02; First posted 2012-02-20 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PaQ™ insulin infusion device (Experimental): PaQ™ insulin infusion device which delivers rapid acting insulin.
  Interventions: Device: PaQ™ insulin infusion device

INTERVENTIONS:
Device: PaQ™ insulin infusion device — Basal/bolus insulin therapy administered by CSII for 4 weeks. First two weeks is transition period to identify correct basal rate for the patient, second 2 weeks is treatment period to evaluate efficacy of CSII device.

SUMMARY:
The purpose of this study is to evaluate the ability of a patient, who has type 2 diabetes (T2DM) who is currently treated with basal/bolus insulin therapy, to use PaQ™ (a simple patch on insulin delivery device) to control his/her blood glucose.

DETAILED DESCRIPTION:
This is a single center, open label, feasibility of use and performance evaluation of PaQ™ (using insulin aspart) in patients with T2DM who are currently receiving basal/bolus insulin therapy with or without oral anti-diabetic drugs (OADs) for glycemic control. The patient's participation in the study is comprised of four phases: screening, baseline evaluation, transition to PaQ™ use, and PaQ™ treatment period. The use of these phases will allow an orderly transition to PaQ™ treatment as well as a reliable construct from which to interpret the final data.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patient's ≥ 30 ≤ 65 years of age.
2. Clinical confirmation of T2DM diagnosis by history and medication usage or glucose tolerance test.
3. Currently treated with insulin using a basal/bolus regimen with or without concurrent use of OADs (metformin and/or glitazone).
4. Currently on a stable insulin regimen "as judged by the investigator" (using an estimate of their basal dose of insulin does not fluctuate by more than ±10% every day) and if he/she is receiving a concurrent oral agent, the dose has remained unchanged for the last 30 days.
5. Currently uses between 20 to 50 units/day basal insulin.

Exclusion Criteria:

1. Uncontrolled hyperglycemia, HbA1c > 9.0% requiring adjustment to his/her insulin regimen.
2. Treated with premixed insulin, or neutral protamine hagedorn (NPH)/glargine/detemir insulin without use of bolus/meal time insulin.
3. Patient has had an episode of severe (assisted) hypoglycemia within the past 30 days.
4. Currently treated with sulfonylurea or incretin-based therapy [glucagon-like peptide-1(GLP-1) agonist or dipeptidyl peptidase-4 (DPP-4) inhibitor].
5. Total daily dose (TDD) of insulin is >100 units/day.
6. Have a meal-time bolus doses that exceeds the capacity of the bolus Insulin Reservoir at any given meal.
7. Have existing dermal irritation on their abdomen or have known hypersensitivity to skin adhesives.
8. Taking or has taken prednisone or cortisone medications in the previous 30 days.
9. Pregnant or is planning to become pregnant during the study period.
10. Has severe medical or psychological condition(s) or chronic conditions/infections that in the opinion of the Investigator would compromise the patient's safety or successful participation in the study.
11. Unable to follow the study clinical investigational plan (CIP)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Patients ability to successfully assemble, fill, prime, apply and use the PaQ™ device | End of two week transition period

SECONDARY OUTCOMES:
Insulin usage | End of two baseline period and end of 2 week treatment period
  Average daily amount of basal insulin and meal time bolus insulin will be calculated
7-point blood glucose reading | Twice per week during baseline period (weeks 1 & 2) and PaQ™ Treatment period (weeks 5 & 6)
  7 - points are pre and 1.5 hours post each meal and at bedtime
Glucose variability | During baseline and PaQ™ treatment period
  Continuous glucose monitoring (CGM) will be performed. Data stored in the CGM will be transferred to a computer at the end of each study period. Glucose variability during each time period will be calculated.
Glucose exposure | During baseline and PaQ™ treatment period
  Continuous glucose monitoring (CGM) will be performed. Data stored in the CGM will be transferred to a computer at the end of each study period. Glucose exposure during each time period will be calculated.
Glucose Stability | During baseline and PaQ™ Treatment Period
  Continuous glucose monitoring (CGM) will be performed. Data stored in the CGM will be transferred to a computer at the end of each study period. Glucose stability during each time period will be calculated.
Infection at cannula insertion site | During transition and PaQ™ treatment period
Occurence of adverse experiences and the number and severity of hypoglycemic episodes | During baseline, transition and PaQ™ treatment period
Quality of Life Questionnaire | At the end of the study
Dermal Irritation | During transition and PaQ™ treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Published in Diabetes Care - Volume 37, May 2014, pages 1476-1479

REFERENCES:
- [Result] Mader JK, Lilly LC, Aberer F, Korsatko S, Strock E, Mazze RS, Damsbo P, Pieber TR. A feasibility study of a 3-day basal-bolus insulin delivery device in individuals with type 2 diabetes. Diabetes Care. 2014 May;37(5):1476-9. doi: 10.2337/dc13-2238. Epub 2014 Mar 5. PMID 24598242